CLINICAL TRIAL: NCT06077929
Title: Evaluation of Variations of Optic Nerve Course in Relation to Posterior Paranasal Sinuses in MDCT at a Tertiary Care Center of Nepal
Brief Title: Optic Nerve Course Variants in Nepali Population
Acronym: ONC
Status: Completed | Type: Observational
Sponsor: Grande International Hospital, Nepal (Other)
Responsible Party: Principal Investigator, PRAJWAL DAHAL, Principal Investigator, Grande International Hospital, Nepal
Other Study IDs: Reg No: 16/2023
Record Dates: First submitted 2023-10-05; First posted 2023-10-11 (Actual); Last update posted 2024-11-07 (Actual); Status verified 2023-10

CONDITIONS: Optic Nerve
Keywords: Optic Nerve Course; De Lano's Classification; Anterior Clinoid Process Pneumatization

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 1 Month
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Rhinosinusitis: Patients with rhinosinusitis
  Interventions: Other: No intervention done

INTERVENTIONS:
Other: No intervention done — No interventions done

SUMMARY:
A retrospective study was conducted on 367 patients. CT PNS and head of the patients were evaluated for type of course of optic nerve according to DeLano's Classification.

DETAILED DESCRIPTION:
A retrospective study was conducted on 367 patients aged 13 years and above. Four investigators, each with 2 to 6 years of experience in the field of radiology, evaluated computed tomography scans of the paranasal sinuses and the head of these patients. The optic nerves were classified into four types based on DeLano's classification, and their respective prevalence rates were determined. Additionally, the prevalence of optic nerve dehiscence and pneumatization of the anterior clinoid process was assessed.

ELIGIBILITY:
Inclusion Criteria: Patients undergoing NCCT PNS and Head for chronic rhinosinusitis, headache and vertigo

Exclusion Criteria:

1. Patient less than 13 years age
2. Patients with recent trauma
3. Patient with large mass/ extensive polyposis

Ages: 13 Years to 94 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Patient of age 13 years and more undergoing NCCT PNS and Head for chronic rhinosinusitis , headache and vertigo
Sampling Method: Probability Sample
Enrollment: 367 (Actual)
Dates: Start 2022-01-01 (Actual); Primary Completion 2023-05-30 (Actual); Study Completion 2023-05-30 (Actual)

PRIMARY OUTCOMES:
Prevalence of different types of optic nerve course | 1.5 years
  Type 4 course is more prevalent than type 3 course

CONTACTS AND LOCATIONS:
Overall Officials: PRAJWAL DAHAL, MD, Principal Investigator — Grande International Hospital
Locations (1):
- Prajwal Dahal, Kathmandu, Bagmati, Nepal

DOCUMENTS (1):
  • Study Protocol (2023-07-30): https://cdn.clinicaltrials.gov/large-docs/29/NCT06077929/Prot_000.pdf